CLINICAL TRIAL: NCT04086641
Title: Functional Assessment of High-profile Crossover Feet in People With Syme's Amputation
Brief Title: Comparison of Prosthetic Feet for People With Syme's Amputation (XF Symes Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Sara Morgan, Assistant Professor, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007788
Record Dates: First submitted 2019-08-16; First posted 2019-09-11 (Actual); Results first posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-11

CONDITIONS: Amputation; Artificial Limb
Keywords: Ankle disarticulation; Syme; Amputation; Prosthesis; Prosthetic foot; Crossover foot; Biomechanics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot 1: Crossover Foot, Foot 2: Energy Storing Foot (Experimental): Participant randomized to crossover foot as first condition, energy storing foot as second condition
  Interventions: Device: Crossover foot; Device: Energy Storing Foot
- Foot 1: Energy Storing Foot, Foot 2: Crossover Foot (Experimental): Participant randomized to energy storing foot as first condition, crossover foot as second condition
  Interventions: Device: Crossover foot; Device: Energy Storing Foot

INTERVENTIONS:
Device: Crossover foot — A prosthetic foot that features an extended strut (keel) that attaches to the posterior proximal aspect of the prosthetic socket.
Device: Energy Storing Foot — A prosthetic foot that features a short strut (keel) that attaches to the distal aspect of the prosthetic socket.

SUMMARY:
The purpose of this study is to compare the functional differences between two types of foot prostheses for people with ankle disarticulation (Syme's) amputations. The two feet being tested are low- and high-profile feet, with the difference being the latter has an extended keel and attaches to the posterior of the prosthetic socket, rather than the distal end. The hypothesis is that the high-profile foot (i.e., the crossover foot) will lead to functional and biomechanical improvements compared to low-profile feet.

DETAILED DESCRIPTION:
Syme's prostheses are typically limited to low-profile prosthetic feet due to clearance restrictions below the prosthetic socket. As a result, the functional benefits provided by the long residual limb are mitigated by prosthetic design limitations. Recently, high-profile, posteriorly-attaching crossover feet have been modified for use with people who have Syme's amputation. Crossover feet theoretically improve motion and energy storage-and-return compared to traditional foot options for the Syme's level. Crossover feet also have the potential to broaden the range of high-impact activities that can be performed with a single prosthesis. However, to date there is no empirical evidence that compares functional differences when walking with high-profile crossover feet compared to low-profile feet for people with Syme's amputation. This mixed-method pilot research will use a randomized, controlled within-participants design. Investigators will assess gait biomechanics, self-reported health outcomes, and qualitative interviews to compare relative advantages and disadvantages of traditional low-profile Syme's feet and high-profile crossover feet. This proposed work will create a foundation for future research that examines the potential benefits of crossover feet in people with Syme's amputation. In addition, results from this research will be used clinically to inform prosthetic options for people with limited clearance for distally-attached prosthetic feet.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Have a unilateral Syme's amputation that occurred >1 year prior
* Owns a crossover foot modified for Syme's use
* Able to walk in the community without assistance
* Able to read and write in English

Exclusion Criteria:

* Have other amputations
* Have a health condition that would limit completion of the study protocol (e.g., skin breakdown, heart disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Morgan, PhD, CPO, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Amplifying Mobility and Performance Laboratory, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Slater C, Hafner BJ, Morgan SJ. Effects of high-profile crossover feet on gait biomechanics in 2 individuals with Syme amputation. Prosthet Orthot Int. 2024 Oct 1;48(5):510-518. doi: 10.1097/PXR.0000000000000295. Epub 2023 Oct 20. PMID 37870369

RESULTS

PARTICIPANT FLOW:
Groups:
- Foot 1: Crossover Foot, Foot 2: Energy Storing Foot: Participants first received a crossover foot, then switched to an energy storing foot. Each foot was utilized for a two week accommodation period at minimum prior to data collection & subsequent switch.
- Foot 1: Energy Storing Foot, Foot 2: Crossover Foot: Participants first received an energy storing foot, then switched to a crossover foot. Each foot was utilized for a two week accommodation period at minimum prior to data collection & subsequent switch.
Period: Foot 1 (Two Week Utilization)
Arm/Group | Foot 1: Crossover Foot, Foot 2: Energy Storing Foot | Foot 1: Energy Storing Foot, Foot 2: Crossover Foot
Started | 2 | 3
Completed | 1 | 1
Not Completed | 1 | 2
Not completed — COVID-19 | 1 | 2
Period: Foot 2 (Two Week Utilization)
Arm/Group | Foot 1: Crossover Foot, Foot 2: Energy Storing Foot | Foot 1: Energy Storing Foot, Foot 2: Crossover Foot
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Foot 1: Crossover Foot, Foot 2: Energy Storing Foot: Participants first received a crossover foot, then switched to an energy storing foot
- Foot 1: Energy Storing Foot, Foot 2: Crossover Foot: Participants first received an energy storing foot, then switched to a crossover foot
- Total: Total of all reporting groups
Arm/Group | Foot 1: Crossover Foot, Foot 2: Energy Storing Foot | Foot 1: Energy Storing Foot, Foot 2: Crossover Foot | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 | 34 | 42.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 0 | 1 | 1
  Canada | 1 | 0 | 1
Amputation Etiology [Count of Participants; unit: Participants]
  Trauma | 1 | 0 | 1
  Cancer | 0 | 1 | 1
MFCL [Count of Participants; unit: Participants] — Medicare Functional Classification Level (K-level) Graded as K-level 0 through 4. K0 indicates the individual does not have the ability or potential to ambulate or transfer safely with or without assistance and a prosthesis does not enhance their quality of life or mobility. The increasing levels indicate higher levels of function, with K4 indicating the individual has the ability or potential for prosthetic ambulation that exceeds basic ambulation skills, exhibiting high impact, stress, or energy levels; typical of the prosthetic demands of the child, active adult, or athlete.
  Participants
    K4 | 1 | 1 | 2
    K1-3 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Ratio Between Sound and Prosthetic Side Step Lengths
Description: The symmetry between prosthetic and sound side step lengths. Step lengths were calculated as the distance between heels from heel strike of the contralateral foot to heel strike of the ipsilateral foot.
Time Frame: Sessions 3 (after 2 weeks of prosthesis 1 wear) and 4 (after 2 weeks of prosthesis 2 wear)
Measure: Number; unit: Sound step length / Pros. step length
Groups:
- Foot 1: Crossover Foot, Foot 2: Energy Storing Foot: First intervention was crossover foot, second was energy storing foot
- Foot 1: Energy Storing Foot, Foot 2: Crossover Foot: First intervention was energy storing foot, second was crossover foot
Arm/Group | Foot 1: Crossover Foot, Foot 2: Energy Storing Foot | Foot 1: Energy Storing Foot, Foot 2: Crossover Foot
Number analyzed (Participants) | 1 | 1
Sound step length / Pros. step length
  Crossover Foot, Slow Walking Speed | 0.88 | 0.87
  Energy Storing Foot, Slow Walking Speed | 1.02 | 0.91
  Crossover Foot, Comfortable Walking Speed | 0.93 | 0.91
  Energy Storing Foot, Comfortable Walking Speed | 0.96 | 0.92
  Crossover Foot, Fast Walking Speed | 0.93 | 0.94
  Energy Storing Foot, Fast Walking Speed | 0.97 | 0.97

2. Primary Outcome: Total Prosthetic Ankle Range of Motion
Description: The change in total angular motion of the ankle in the sagittal plane (e.g., dorsiflexion & plantarflexion) during stance phase between prosthetic feet, in degrees
Time Frame: Sessions 3 (after 2 weeks of prosthesis 1 wear) and 4 (after 2 weeks of prosthesis 2 wear)
Measure: Number; unit: degrees
Arm/Group | Foot 1: Crossover Foot, Foot 2: Energy Storing Foot | Foot 1: Energy Storing Foot, Foot 2: Crossover Foot
Number analyzed (Participants) | 1 | 1
degrees
  Crossover Foot, Slow Walking Speed | 14.04 | 14.20
  Energy Storing Foot, Slow Walking Speed | 7.94 | 9.03
  Crossover Foot, Comfortable Walking Speed | 17.91 | 16.24
  Energy Storing Foot, Comfortable Walking Speed | 11.17 | 9.63
  Crossover Foot, Fast Walking Speed | 16.74 | 17.53
  Energy Storing Foot, Fast Walking Speed | 11.91 | 11.20

3. Primary Outcome: Prosthetic-side Energy Return
Description: Intersegmental flow of power out of the prosthesis
Time Frame: Sessions 3 (after 2 weeks of prosthesis 1 wear) and 4 (after 2 weeks of prosthesis 2 wear)
Measure: Number; unit: W/kg
Arm/Group | Foot 1: Crossover Foot, Foot 2: Energy Storing Foot | Foot 1: Energy Storing Foot, Foot 2: Crossover Foot
Number analyzed (Participants) | 1 | 1
W/kg
  Crossover Foot, Slow Walking Speed | 0.86 | 1.27
  Energy Storing Foot, Slow Walking Speed | 0.32 | 0.36
  Crossover Foot, Comfortable Walking Speed | 2.18 | 2.32
  Energy Storing Foot, Comfortable Walking Speed | 0.90 | 0.53
  Crossover Foot, Fast Walking Speed | 2.82 | 4.22
  Energy Storing Foot, Fast Walking Speed | 1.53 | 0.75

4. Primary Outcome: Peak Sound-side Limb Loading
Description: Maximum vertical ground reaction force in early stance
Time Frame: Sessions 3 (after 2 weeks of prosthesis 1 wear) and 4 (after 2 weeks of prosthesis 2 wear)
Measure: Number; unit: Ratio (Newtons/body weight)
Arm/Group | Foot 1: Crossover Foot, Foot 2: Energy Storing Foot | Foot 1: Energy Storing Foot, Foot 2: Crossover Foot
Number analyzed (Participants) | 1 | 1
Ratio (Newtons/body weight)
  Crossover Foot, Slow Walking Speed | 1.06 | 1.04
  Energy Storing Foot, Slow Walking Speed | 1.06 | 1.16
  Crossover Foot, Comfortable Walking Speed | 1.07 | 1.17
  Energy Storing Foot, Comfortable Walking Speed | 1.23 | 1.29
  Crossover Foot, Fast Walking Speed | 1.37 | 1.53
  Energy Storing Foot, Fast Walking Speed | 1.43 | 1.45

5. Secondary Outcome: Preference Questionnaire
Description: At the end of the study, participants will engage in a preference questionnaire with open-ended follow-up questions to elicit preferences and experiences with both feet. Questions will ask about overall preference, and preference for a range of mobility activities (e.g., "Which foot did you prefer overall, and why?" and "Which foot did you prefer for walking up stairs, and why?").
Time Frame: Session 4 (after 4 weeks of prosthesis wear, 2 weeks of prosthesis 1 and 2 weeks of prosthesis 2)
Measure: Count of Participants; unit: Participants
Arm/Group | Foot 1: Crossover Foot, Foot 2: Energy Storing Foot | Foot 1: Energy Storing Foot, Foot 2: Crossover Foot
Number analyzed (Participants) | 1 | 1
Participants
  Walking on inclines: Prefers Crossover Foot | 1 | 1
  Walking on inclines: Prefers Energy Storing Foot | 0 | 0
  Walking on inclines: No preference | 0 | 0
  Walking on inclines: Not applicable | 0 | 0
  Walking on declines: Prefers Crossover Foot | 1 | 0
  Walking on declines: Prefers Energy Storing Foot | 0 | 0
  Walking on declines: No preference | 0 | 1
  Walking on declines: Not applicable | 0 | 0
  Ascending stairs: Prefers Crossover Foot | 1 | 1
  Ascending stairs: Prefers Energy Storing Foot | 0 | 0
  Ascending stairs: No preference | 0 | 0
  Ascending stairs: Not applicable | 0 | 0
  Descending stairs: Prefers Crossover Foot | 1 | 1
  Descending stairs: Prefers Energy Storing Foot | 0 | 0
  Descending stairs: No preference | 0 | 0
  Descending stairs: Not applicable | 0 | 0
  Walking slowly: Prefers Crossover Foot | 0 | 1
  Walking slowly: Prefers Energy Storing Foot | 0 | 0
  Walking slowly: No preference | 1 | 0
  Walking slowly: Not applicable | 0 | 0
  Walking quickly: Prefers Crossover Foot | 1 | 1
  Walking quickly: Prefers Energy Storing Foot | 0 | 0
  Walking quickly: No preference | 0 | 0
  Walking quickly: Not applicable | 0 | 0
  Running: Prefers Crossover Foot | 1 | 1
  Running: Prefers Energy Storing Foot | 0 | 0
  Running: No preference | 0 | 0
  Running: Not applicable | 0 | 0
  Walking over uneven terrain: Prefers Crossover Foot | 0 | 1
  Walking over uneven terrain: Prefers Energy Storing Foot | 0 | 0
  Walking over uneven terrain: No preference | 1 | 0
  Walking over uneven terrain: Not applicable | 0 | 0
  Standing up from a chair: Prefers Crossover Foot | 1 | 0
  Standing up from a chair: Prefers Energy Storing Foot | 0 | 0
  Standing up from a chair: No preference | 0 | 1
  Standing up from a chair: Not applicable | 0 | 0
  Sitting down in a chair: Prefers Crossover Foot | 0 | 0
  Sitting down in a chair: Prefers Energy Storing Foot | 0 | 0
  Sitting down in a chair: No preference | 1 | 1
  Sitting down in a chair: Not applicable | 0 | 0
  Turning on the prosthetic side: Prefers Crossover Foot | 1 | 1
  Turning on the prosthetic side: Prefers Energy Storing Foot | 0 | 0
  Turning on the prosthetic side: No preference | 0 | 0
  Turning on the prosthetic side: Not applicable | 0 | 0
  Getting in and out of a car: Prefers Crossover Foot | 0 | 1
  Getting in and out of a car: Prefers Energy Storing Foot | 0 | 0
  Getting in and out of a car: No preference | 1 | 0
  Getting in and out of a car: Not applicable | 0 | 0
  Playing sports: Prefers Crossover Foot | 1 | 1
  Playing sports: Prefers Energy Storing Foot | 0 | 0
  Playing sports: No preference | 0 | 0
  Playing sports: Not applicable | 0 | 0
  Standing for long periods: Prefers Crossover Foot | 0 | 1
  Standing for long periods: Prefers Energy Storing Foot | 0 | 0
  Standing for long periods: No preference | 1 | 0
  Standing for long periods: Not applicable | 0 | 0
  Walking in sand: Prefers Crossover Foot | 0 | 0
  Walking in sand: Prefers Energy Storing Foot | 0 | 1
  Walking in sand: No preference | 0 | 0
  Walking in sand: Not applicable | 1 | 0
  Walking when you can't see your feet: Prefers Crossover Foot | 0 | 1
  Walking when you can't see your feet: Prefers Energy Storing Foot | 0 | 0
  Walking when you can't see your feet: No preference | 1 | 0
  Walking when you can't see your feet: Not applicable | 0 | 0
  Walking when carrying a heavy load: Prefers Crossover Foot | 0 | 1
  Walking when carrying a heavy load: Prefers Energy Storing Foot | 0 | 0
  Walking when carrying a heavy load: No preference | 1 | 0
  Walking when carrying a heavy load: Not applicable | 0 | 0
  Walking in small spaces: Prefers Crossover Foot | 0 | 1
  Walking in small spaces: Prefers Energy Storing Foot | 0 | 0
  Walking in small spaces: No preference | 1 | 0
  Walking in small spaces: Not applicable | 0 | 0
  Dancing: Prefers Crossover Foot | 1 | 1
  Dancing: Prefers Energy Storing Foot | 0 | 0
  Dancing: No preference | 0 | 0
  Dancing: Not applicable | 0 | 0
  Riding a bicycle: Prefers Crossover Foot | 0 | 1
  Riding a bicycle: Prefers Energy Storing Foot | 0 | 0
  Riding a bicycle: No preference | 1 | 0
  Riding a bicycle: Not applicable | 0 | 0

6. Secondary Outcome: Change in Prosthetic Limb Users Survey of Mobility (PLUS-M) 12-item Short Form Version 1.2
Description: Self-reported measure of mobility, the PLUS-M 12-item Short Form is a single measure, scores range from 17.5-76.6, higher scores represent better mobility.
Time Frame: Sessions 3 (after 2 weeks of prosthesis 1 wear) and 4 (after 2 weeks of prosthesis 2 wear)
Measure: Number; unit: score on a scale
Arm/Group | Foot 1: Crossover Foot, Foot 2: Energy Storing Foot | Foot 1: Energy Storing Foot, Foot 2: Crossover Foot
Number analyzed (Participants) | 1 | 1
score on a scale
  Crossover Foot | 64.5 | 71.4
  Energy Storing Foot | 64.5 | 62.5

7. Secondary Outcome: Change in Activities-Specific Balance Confidence Scale (ABC)
Description: Self-reported measure of balance confidence, the ABC is a single measure, scores range from 0-4, higher scores represent better balance confidence.
Time Frame: Sessions 3 (after 2 weeks of prosthesis 1 wear) and 4 (after 2 weeks of prosthesis 2 wear)
Measure: Number; unit: score on a scale
Arm/Group | Foot 1: Crossover Foot, Foot 2: Energy Storing Foot | Foot 1: Energy Storing Foot, Foot 2: Crossover Foot
Number analyzed (Participants) | 1 | 1
score on a scale
  Crossover Foot | 3.53 | 4
  Energy Storing Foot | 3.63 | 4

8. Secondary Outcome: Change in Trinity Amputation and Prosthesis Experience Scales- Revised Aesthetic Satisfaction
Description: Self-reported measures of aesthetic prosthetic satisfaction, scores on items are averaged and range from 0-2, higher values represent more satisfaction (better outcome)
Time Frame: Sessions 3 (after 2 weeks of prosthesis 1 wear) and 4 (after 2 weeks of prosthesis 2 wear)
Measure: Number; unit: score on a scale
Arm/Group | Foot 1: Crossover Foot, Foot 2: Energy Storing Foot | Foot 1: Energy Storing Foot, Foot 2: Crossover Foot
Number analyzed (Participants) | 1 | 1
score on a scale
  Crossover Foot | 0.33 | 2
  Energy Storing Foot | 1 | 1

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year
Description: At each research session, a Physical Health questionnaire was administered in which participants reported other non-serious adverse events relevant to the study, including residual limb sores, phantom pain, and loss of sensation or numbness in residual limb.
Groups:
- Foot 1: Crossover Foot, Foot 2: Energy Storing Foot: Participants first received the crossover foot, then switched to the energy storing
- Foot 1: Energy Storing Foot, Foot 2: Crossover Foot: Participants first received the energy storing foot, then switched to the crossover foot
Arm/Group | Foot 1: Crossover Foot, Foot 2: Energy Storing Foot | Foot 1: Energy Storing Foot, Foot 2: Crossover Foot
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Small clinical population & resultant study sample size, disallowing inferential statistical analysis; COVID-19 pandemic resulting in cessation of human subjects research prior to obtaining data on all enrolled subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT04086641/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT04086641/SAP_001.pdf